CLINICAL TRIAL: NCT01327209
Title: Blood Glucose Monitoring System Clinical Study
Acronym: BGMS
Status: Completed | Type: Observational
Sponsor: Intuity Medical, Inc (Industry)
Responsible Party: Dr. Richard Bergenstal, International Diabetes Center
Other Study IDs: TP-0000145
Record Dates: First submitted 2011-03-30; First posted 2011-04-01 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with diabetes

SUMMARY:
Verify the following with blood glucose monitoring system:

* precision and accuracy versus YSI reference
* user evaluation
* labeling comprehension

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with Diabetes
* Be between 12 and 70 years of age
* Be able to read, write, and understand English
* Be able and willing to give Informed Consent
* Have used an SMBG meter system for at least one year
* Be currently testing blood glucose levels at least once per day

Exclusion Criteria:

* Inability to provide Informed Consent
* Subject does not meet Inclusion Criteria
* Subject does not agree to test for infectious diseases per clinical protocol
* Subject has minimally one positive test for any infectious disease listed under Exclusion Criteria per protocol
* Subject with any condition (in addition to those which are listed in the pre-screen Exclusion Criteria tests) which in the opinion of the Investigator may place the subject or site personnel at excessive risk
* Subject's physical condition/limitation prevents the person from using a BGMS on their own

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People who have been diagnosed with diabetes and are testing their blood glucose level at least once per day.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2010-12; Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bergenstal, MD, Principal Investigator — Park Nicollett Institue - International Diabetes Center
Locations (4):
- United States (4):
  - University of San Diego, San Diego, California
  - University of Miami - School of Medicine, Miami, Florida
  - Park Nicollett Institute - International Diabetes Center, Minneapolis, Minnesota
  - Cetero Research DGD, San Antonio, Texas